CLINICAL TRIAL: NCT06347679
Title: Effects of Aromatherapy on Anxiety and Pain During Dental Treatment in Adults: a Randomized Controlled Clinical Trial
Brief Title: Effects of Aromatherapy on Anxiety and Pain During Dental Treatment in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, He Cai, Assistant Researcher, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WCHSIRB-CT-2024-160
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: single-note sweet orange essential oil (Experimental)
  Interventions: Other: Aroma diffuser with single-note sweet orange essential oil
- Group 2: single-note tea tree essential oil (Experimental)
  Interventions: Other: Aroma diffuser with single-note tea tree essential oil
- Group 3: water (Sham Comparator)
  Interventions: Other: Aroma diffuser with water

INTERVENTIONS:
Other: Aroma diffuser with single-note sweet orange essential oil — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of 100% concentration single-note sweet orange essential oil into the aroma diffuser reservoir containing 120 ml of water.
  Arms: Group 1: single-note sweet orange essential oil
Other: Aroma diffuser with single-note tea tree essential oil — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of 100% concentration single-note tea tree essential oil into the aroma diffuser reservoir containing 120 ml of water.
  Arms: Group 2: single-note tea tree essential oil
Other: Aroma diffuser with water — In a space of 3*4*2.6 cubic meters, positioned 10 cm away from the patient, add 4-6 drops (each drop being 0.05 ml) of water into the aroma diffuser reservoir containing 120 ml of water.
  Arms: Group 3: water

SUMMARY:
Dental anxiety is a common problem in dental care. The aim of this protocol is to evaluate the effect of orange and tea essential oil for the control of anxiety and pain in adults during dental treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need dental treatment, such as resin filling, root canal treatment, periodontal initial treatment, tooth extraction, etc.
* Be able to understand the purpose of the study and volunteer to take part in the study.
* Be able to complete all assessments and follow-up during the study.

Exclusion Criteria:

* Patients who are allergic to the ingredients of the essential oils used in the experiment or to the materials used in the dental treatment.
* Patients who underwent only an oral examination.
* Patients with severe heart disease, hypertension, respiratory disease, or other systemic conditions that were not eligible for trial participation.
* Pregnant or lactating women.
* People with depressive symptoms, anxiety disorders or other mental illnesses that affect their mood state.
* People who are using sedative or analgesic drugs.
* Recent or current users of essential oil.
* Any circumstances considered by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety scale 1 - Modified Dental Anxiety Scale (MDAS) | 5 minutes before operation/during operation (immediately after the most painful procedure)/immediately after operation
  The Modified Dental Anxiety Scale (MDAS) consists of 4 questions each with a 5 category rating scale, ranging from 'not anxious' to 'extremely anxious', hence, the total score varies from 4 to 20, with higher obtained scores describing more elevated levels of dental anxiety. MDAS is recorded before, during and after operation.
Pain scale - Visual Analog Scale (VAS) | 5 minutes before operation/during operation (immediately after the most painful procedure)/immediately after operation
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." VAS is recorded before, during and after operation.

SECONDARY OUTCOMES:
Anxiety scale 2 - State-Trait Anxiety Inventory for State Anxiety (STAI-S) | 5 minutes before operation/ immediately after operation
  The STAI-S evaluates the subjective feelings of tension, worry, nervousness, apprehension, and autonomic nervous system activation. This self-completed inventory consisted of 20 items on a four-point Likert scale running from one (i.e., not at all) to four (i.e., very much). Hence, the total score varies from 20 to 80, with higher obtained scores describing more elevated levels of anxiety. STAI-S is recorded before and after operation,
Vital sign 1 - systolic blood pressure (SBP) | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation
  systolic blood pressure (SBP) is measured using a manual sphygmomanometer, before, during and after operation.
Vital sign 2 - diastolic blood pressure (DBP) | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation
  diastolic blood pressure (DBP) is measured using a manual sphygmomanometer, before, during and after operation.
Vital sign 3 - heart rate (HR） | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation
  Heart rate (HR）is measured as pulse rate using an oximeter, before, during and after operation.
Vital sign 4 - oxygen saturation (SpO2） | 5 minutes before operation/during operation (immediately after the most painful procedure, and every 10min after)/immediately after operation
  oxygen saturation (SpO2）is measured using an oximeter, before, during and after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology SIchuan University, Chengdu, Sichuan, China